CLINICAL TRIAL: NCT05165706
Title: Longitudinal Multi-Omic Profiles to Reveal Mechanisms of Obesity-Mediated Insulin Resistance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Tracey McLaughlin, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 40195; 5R01DK110186-02 (NIH)
Record Dates: First submitted 2018-07-03; First posted 2021-12-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes; Insulin Resistance; Obesity; Nonalcoholic Steatohepatitis; Nonalcoholic Fatty Liver; Diet Modification
Keywords: Metabolomics; Low Fat Diet; Low Carbohydrate Diet; Microbiome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Insulin Resistance; Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediterranean Low Carbohydrate Diet (Experimental): Assigned participants will receive instruction by a registered dietitian on a diet that is high in unsaturated fats and low in carbohydrates. Total caloric intake will be adjusted to induce a supervised metabolic challenge defined as weight gain of approximately 2.5 kg over 5 weeks followed by 3-5kg weight loss over 8 weeks.
  Interventions: Behavioral: Dietary Intervention Mediterranean Low Carbohydrate Diet
- Standard Low Carbohydrate Diet (Experimental): Assigned participants will receive instruction by a registered dietitian on a low carbohydrate diet that is high in fats found in the typical American diet. Total caloric intake will be adjusted to induce a supervised metabolic challenge defined as weight gain of approximately 2.5 kg over 5 weeks followed by 3-5kg weight loss over 8 weeks.
  Interventions: Behavioral: Dietary Intervention Standard Low Carbohydrate Diet
- Low Fat, Healthy Carbohydrate Diet (Experimental): Assigned participants will receive instruction by a registered dietitian on a low fat diet that is high in complex carbohydrates. Total caloric intake will be adjusted to induce a supervised metabolic challenge defined as weight gain of approximately 2.5 kg over 5 weeks followed by 3-5kg weight loss over 8 weeks.
  Interventions: Behavioral: Dietary Intervention Standard Low Fat Diet

INTERVENTIONS:
Behavioral: Dietary Intervention Mediterranean Low Carbohydrate Diet — Assigned participants will receive instruction by a registered dietitian on a diet that is high in unsaturated fats and low in carbohydrates. Total caloric intake will be adjusted to induce a supervised metabolic challenge defined as weight gain of approximately 2.5 kg over 5 weeks followed by 3-5kg weight loss over 8 weeks.
  Arms: Mediterranean Low Carbohydrate Diet
Behavioral: Dietary Intervention Standard Low Carbohydrate Diet — Assigned participants will receive instruction by a registered dietitian on a low carbohydrate diet that is high in fats found in the typical American diet. Total caloric intake will be adjusted to induce a supervised metabolic challenge defined as weight gain of approximately 2.5 kg over 5 weeks followed by 3-5kg weight loss over 8 weeks.
  Arms: Standard Low Carbohydrate Diet
Behavioral: Dietary Intervention Standard Low Fat Diet — Assigned participants will receive instruction by a registered dietitian on a low fat diet that is high in complex carbohydrates. Total caloric intake will be adjusted to induce a supervised metabolic challenge defined as weight gain of approximately 2.5 kg over 5 weeks followed by 3-5kg weight loss over 8 weeks.
  Arms: Low Fat, Healthy Carbohydrate Diet

SUMMARY:
This 12-week controlled diet and weight intervention study seeks to define the molecular pathways that link excess body weight to the development of insulin resistance (IR). Blood, adipose and stool are sampled at three timepoints; baseline, peak weight (4 weeks) and post weight loss to monitor changes in cellular processes. Additionally, direct insulin sensitivity testing, and radiological measurement of visceral fat and intrahepatic fat content is measured at three timepoints to correlate clinical indices with cellular changes.

DETAILED DESCRIPTION:
Obesity has become an epidemic worldwide. Metabolic/cardiovascular complications of obesity are likely related to the fact that obese individuals tend to be insulin resistant (IR). While insulin- mediated glucose uptake (IMGU) correlates with adipose tissue mass, not all obese individuals are IR, and metabolic and cardiovascular profiles of those who are IR vs insulin sensitive (IS) differ significantly. Why one individual who reaches a BMI of 30 kg/m2 will develop IR and another with similar BMI and activity level remains IS is unclear. Furthermore, while insulin sensitivity improves with weight loss, this response varies as well. Given that fat mass per se does not fully explain the obesity contribution to IMGU, itis likely that differential adipocyte function plays a role. With this study, our purpose is to employ an integrated omics strategy to identify analyte/pathway signatures in blood and adipose tissue that characterize IR versus IS states and expand our biological knowledge of the mechanisms underlying IR.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-65
* BMI 25-35 kg/m2
* Stable body weight
* Nondiabetic

Exclusion Criteria:

Patients with;

* diabetes
* major organ disease
* history of liposuction or bariatric surgery
* active eating or psychiatric disorder
* pregnancy or lactation, heavy alcohol use
* recent change in weight (over the past 12 weeks)
* use of weight loss medication, statins, or oral steroids

Clinical screening exclusions;

* hematocrit < 33%
* fasting glucose >/= 126 mg/dL
* blood pressure >160/100 mmHg

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-01-31 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the 2-stage Steady State Plasma Glucose test | Peak weight (4 weeks)
  Compare direct measurement of insulin sensitivity after 4 week diet and weight intervention
Change from baseline on the radiographic measurement of visceral to subcutaneous (V:S) fat ratio | Peak weight (4 weeks)
  Compare measurement of abdominal V:S fat volume via computed tomography (CT) after 4 week diet and weight intervention
Change from baseline on the magnetic-resonance based measurement of intrahepatic lipid deposition | Peak weight (4 weeks)
  Compare measurement of liver fat content via magnetic resonance spectroscopy (MRS) after 4 week diet and weight intervention
Change from peak weight on the 2-stage Steady State Plasma Glucose test | Post-weight loss (8 weeks)
  Compare direct measurement of insulin sensitivity after 8 week diet and weight intervention
Change from baseline on the radiographic measurement of visceral to subcutaneous (V:S) fat ratio | Post-weight loss (8 weeks)
  Compare measurement of abdominal V:S fat volume via computed tomography (CT) after 8 week diet and weight intervention
Change from baseline on the magnetic-resonance based measurement of intrahepatic lipid deposition | Post-weight loss (8 weeks)
  Compare measurement of liver fat content via magnetic resonance spectroscopy (MRS) after 8 week diet and weight intervention
Measurement of markers of lipid and carbohydrate metabolism and inflammation from adipose mRNA | Baseline
  Compare adipose tissue transcripts such as known MODY transcription factors, defensin chemokine receptors, and platelet activation factors measured by PCR between participants identified as Insulin sensitive (IS) and Insulin resistant (IR) using the 2-stage Steady State Plasma Glucose test.
Quantification of plasma inflammatory cytokine levels in serum samples by Luminex immunoassay | Baseline
  Compare plasma inflammatory cytokine levels in serum samples as measured by Luminex immunoassay between participants identified as Insulin Sensitive (IS) and Insulin Resistant (IR) using the 2-stage Steady State Plasma Glucose test.
Change from baseline in plasma inflammatory cytokine levels in serum samples as measured by Luminex immunoassay | Peak Weight (4 weeks)
  Compare intra-personal levels of plasma inflammatory cytokines as measured by Luminex immunoassay after 4 week diet and weight intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MD, Principal Investigator — Stanford University, Department of Medicine, Division of Endocrinology
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No